CLINICAL TRIAL: NCT00585364
Title: SCCOR in Host Factors in Chronic Lung Diseases: Mechanisms of Immune Tolerance and Inflammation in Allergic Bronchopulmonary Aspergillosis (ABPA) in Patients With Cystic Fibrosis
Brief Title: Mechanisms of Immune Tolerance and Inflammation in Patients With Cystic Fibrosis With ABPA
Acronym: ABPA
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jay Kolls, PI, University of Pittsburgh
Other Study IDs: SCCOR; P50HL084932 (NIH)
Record Dates: First submitted 2008-01-01; First posted 2008-01-03 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Cystic Fibrosis; Allergic Bronchopulmonary Aspergillosis
Keywords: Allergic Bronchopulmonary Aspergillosis; Aspergillus fumigatus; cytokine expression
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The CF subject's blood will be processed to establish a cell line (lymphocyte transformation) for a source of DNA for future genetic studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CF (non-ABPA): cystic fibrosis and culture positive for A. fumigatus in airway cultures.
- CF and ABPA: cystic fibrosis and diagnosis of ABPA
- healthy control: healthy non-CF

SUMMARY:
The goal of this study is to identify the immunological factors that influence a patient's response to the presence of the fungus Aspergillus fumigatus (A. fumigatus) in the lungs. In patients with cystic fibrosis (CF), this fungus is not known to cause damage to the lungs, but some patients respond with an allergic reaction that may cause wheeze, cough, or difficulty breathing. Approximately 230 patients will be enrolled with an additional 60 people who do not have CF and who do not have a history of asthma to serve as a comparison group.

DETAILED DESCRIPTION:
In this cohort the investigators will study blood T-cell responses to Aspergillus antigens to determine if patients with ABPA have greater type 2 responses as measured by IL-13 compared to CF or non-CF controls.

ELIGIBILITY:
Inclusion Criteria:

(CF)

* diagnosis of CF
* age 6 years or older
* presence of A. fumigatus in culture of airway flora, or the presence of one or more of the diagnostic criteria for ABPA (Control)
* age and sex matched to CF population

Exclusion Criteria:

(CF)

* uncontrolled CF-related diabetes mellitus
* use of oral steroids at a dose ≥ 0.5 mg/kg/day
* history of lung transplantation
* pulmonary exacerbation as defined by requirement for use of intravenous antibiotics or need for hospitalization within the preceding 14 days.
* patients who have a diagnosis of HIV and have a CD4+ Tcell count below 500 cells/ml will be excluded (control)
* asthma

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects with CF who have A. fumigatus in cultures of airway flora and receive clinical care at the Antonio J. and Janet Palumbo Cystic Fibrosis Center at Children's Hospital of Pittsburgh. Age (± 1 year) and sex matched healthy, non CF controls will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2005-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that the white blood cells of CF patients with ABPA will demonstrate increased inflammatory cytokine expression in response to binding of A. fumigatus antigens compared to white blood cells from non-ABPA patients. | baseline, 6 month follow-up, ABPA exacerbation

SECONDARY OUTCOMES:
To test the hypothesis that T cells from CF patients with ABPA will have decreased adaptive regulatory function | baseline, 6 month follow-up, ABPA exacerbation
To test the hypothesis that surface-bound TGF beta is critical for the development and maintenance of immune tolerance to A. fumigatus antigens | baseline, 6 month follow-up, ABPA exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Jay K Kolls, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This was an observational trial that involved no device or drug.